CLINICAL TRIAL: NCT07152756
Title: Impact of a One-Week Discontinuation of Semaglutide on Gastric Retention and Endoscopic Mucosal Visibility Scores: A Single-Center, Prospective, Observational Study
Brief Title: Impact of a One-Week Discontinuation of Semaglutide on Gastric Retention and Endoscopic Mucosal Visibility Scores
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: 2025K248
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Gastric Retention
Keywords: Semaglutide; Gastric Retention; Esophagogastroduodenoscopy
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: one-week discontinuation of semaglutide before EGD
  Interventions: Procedure: Esophagogastroduodenoscopy
- non-exposure group: no semaglutide use before EGD
  Interventions: Procedure: Esophagogastroduodenoscopy

INTERVENTIONS:
Procedure: Esophagogastroduodenoscopy — Assess the gastric retention and the endoscopic mucosal visibility score during esophagogastroduodenoscopy

SUMMARY:
A prospective, single-center, observational study to compare the risk of gastric retention and endoscopic mucosal visibility between the exposure group (one-week discontinuation of semaglutide before EGD) and non-exposure group (no semaglutide use before EGD)

DETAILED DESCRIPTION:
Glucagon-like peptide-1 receptor agonists (GLP-1RAs) mimic the action of endogenous GLP-1 hormones by activating GLP-1 receptors in the pancreas, brain, and gastrointestinal tract. This results in enhanced insulin secretion, suppressed glucagon release, delayed gastric emptying, and improved glycemic control and weight management in patients with type 2 diabetes. However, this pharmacological mechanism also increases the risk of gastric retention.

Multiple previous studies and recent meta-analyses have demonstrated that continued use of GLP-1RAs is associated with an elevated risk of gastric retention, which may lead to aspiration and significantly increase the risks associated with anesthesia. As a result, several recent expert consensus statements and clinical guidelines-including the 2023 ASA Expert Consensus and the 2025 ASGE Clinical Guidelines-recommend withholding weekly GLP-1RA agents for at least one week prior to procedures requiring anesthesia, regardless of dosage. For patients whose discontinuation period is less than one week, preoperative gastric ultrasound is advised to rule out gastric retention before proceeding with anesthesia; otherwise, anesthesia should be administered as for a "full stomach".

However, both the ASA consensus and ASGE guidelines acknowledge that clinical evidence supporting the effectiveness of a one-week GLP-1RA discontinuation in reducing gastric retention remains insufficient. A recent retrospective study reported that the risk of gastric retention remained significantly elevated even after one week of discontinuation compared to non-users. Only after a two-week discontinuation and in the absence of gastrointestinal symptoms such as bloating, nausea, or vomiting did the gastric retention risk return to normal levels.

Taken together, the current recommendation of a one-week discontinuation before anesthesia for weekly GLP-1RAs remains open to improvement and warrants further investigation through high-quality clinical studies to determine the optimal discontinuation interval.

In this study, we propose a single-center, prospective, observational study focusing on semaglutide, the most widely used weekly GLP-1RA. Individuals who have discontinued semaglutide for one week prior to undergoing painless endoscopy (with the last dose administered 8-14 days before the procedure) will be enrolled as the exposure group. Those who have not used any GLP-1RAs prior to the procedure will serve as the non-exposure group. The study aims to compare the risk of gastric retention and the endoscopic mucosal visibility score between the two groups, in order to explore the most appropriate semaglutide discontinuation interval before painless endoscopy.

ELIGIBILITY:
Inclusion Criteria

1. Subjects who have either: (i) been on long-term semaglutide therapy (≥4 weeks, any dosage) and discontinued use for one week prior to gastroscopy (with the last dose 8-14 days before the procedure), or(ii) never used semaglutide.
2. For patients with diabetes mellitus (DM), HbA1c < 9% to ensure adequate glycemic control.
3. Age ≥ 18 years, with no restriction on sex.
4. American Society of Anesthesiologists (ASA) physical status classification I-II.
5. Fasting for at least 8 hours and no water intake for at least 4 hours before gastroscopy.
6. Undergoing painless (sedated) endoscopy.

Exclusion Criteria

1. History of hiatal hernia or any previous gastric surgery (including gastrectomy, Roux-en-Y gastric bypass, etc.).
2. Pregnancy.
3. Medically unfit for gastrointestinal endoscopy.
4. Deemed unsuitable for participation at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing sedated endoscopy who had discontinued semaglutide for one week prior to the procedure (with the last dose administered 8-14 days before EGD) were assigned to the exposure group, while those who had not used semaglutide were assigned to the non-exposure group.
Sampling Method: Probability Sample
Enrollment: 418 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of gastric retention | immediately after the esophagogastroduodenoscopy
  Gastric retention was defined as the presence of solid residues in the stomach or liquid retention exceeding 1.5 mL/kg

SECONDARY OUTCOMES:
Gastric Mucosal Visibility Score | immediately after the esophagogastroduodenoscopy
Rate of hypoxemia and aspiration events | immediately after the esophagogastroduodenoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)